CLINICAL TRIAL: NCT03846414
Title: Real World Study of PEGylated Recombinant Human Granulocyte Stimulating Factor(PEG-rhG-CSF) in Prevention of Chemotherapy-induced Neutropenia
Brief Title: Real World Study of PEG-rhG-CSF in Prevention of Chemotherapy-induced Neutropenia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSPC-JYL-RWS-07
Record Dates: First submitted 2019-02-14; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Chemotherapy-induced Neutropenia; Myelosuppression
Keywords: PEG-rhG-CSF; Pegfilgrastim
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEG-rhG-CSF group: This group comprised 1000 patients who received a single subcutaneous injection of PEG-rhG-CSF 24 hours after the end of chemotherapy for each chemotherapy cycle. The dose of PEG-rhG-CSF is determined by the patients' body weight, patients with body weight ≥45 kg is given to PEG-rhG-CSF 6 mg each time, patients<45 kg is given to PEG-rhG-CSF 3 mg each time.
  Interventions: Drug: PEG-rhG-CSF
- rhG-CSF group: This group comprised 500 patients who received rhG-CSF 5 μg/kg/day by subcutaneous injection 24 hours after the end of chemotherapy or the appearance of CIN until the ANC was ≥2.0x109/L for each chemotherapy cycle.

INTERVENTIONS:
Drug: PEG-rhG-CSF — PEG-rhG-CSF was administered 24 hours after the end of chemotherapy for each chemotherapy cycle.
  Other Names: Jinyouli
  Groups: PEG-rhG-CSF group

SUMMARY:
The aim of this study is to observe and evaluate the cost-effectiveness,efficacy and safety of PEG-rhG-CSF in preventing chemotherapy-induced neutropenia(CIN) of cancer patients in the real world.1000 patients with non-myeloid malignancy who is planned to receive PEG-rhG-CSF for CIN prevention and 500 patients with non-myeloid malignancy who is planned to receive rhG-CSF for CIN prevention or treatment were prospectively recruited.The primary outcome was cost-effectiveness and second outcome was febrile neutropenia,the incidence and duration of grade IV neutropenia,chemotherapy delay,incidence of reduced dose of chemotherapy and relative dose intensity of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age≥18 years old, male or female
2. Diagnosis of non-myeloid malignant solid tumors
3. Patients are planned to perform chemotherapy and preventive use the PEG-rhG-CSF or preventive or therapeutic use of rhG-CSF after chemotherapy
4. Patients' mental status are well, could understand the study and willing to participate the study, sign the informed consent form
5. The investigator believes that patients can benefit from this study

Exclusion Criteria:

1. Patients who have been confirmed to be allergic to Jinyouli® or rhG-CSF or its excipients
2. Pregnant or lactating women and women who plan to be pregnant during clinical observation
3. Other patients that the doctor believe not suitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 patients with non-myeloid malignancy who is planned to receive PEG-rhG-CSF for CIN prevention and 500 patients with non-myeloid malignancy who is planned to receive rhG-CSF for CIN prevention or treatment were prospectively recruited.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-02-13 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Cost-Effectiveness | through the chemotherapy cycles of PEG-rhG-CSF or rhG-CSF treatment,an average of 3 month
  Based on the results of the incidence of febrile neutropenia(FN) and the cost perFN in each group, the incremental cost-effectiveness ratio were estimated using the following formula: (CostA-CostB)/(OutcomeA-OutcomeB)

SECONDARY OUTCOMES:
The incidence of febrile neutropenia | From date of randomization until the date of the study completion,an average of 3 month
  Febrile neutropenia (FN) is defined as oral temperature >38.3 ℃(under arm temperature >38.1 ℃) or continuous measurement of oral temperature >38℃(under arm temperature >37.8℃) in 2h, and absolute neutrophil count(ANC) <0.5×10^9/L, or expected to be <0.5×10^9/L
The incidence of grade IV neutropenia | From date of randomization until the date of the study completion,an average of 3 month
  Grade IV neutropenia is defined as the absolute neutrophil count(ANC)<0.5×10^9/L
The duration of grade IV neutropenia in every chemotherapy cycle | From date of randomization until the date of the study completion,an average of 3 month
  Defined as days when the ANC<2.0×10^9/L occurs to the time when the ANC≥2.0×10^9/L, take the median
The incidence of the chemotherapy delay | From date of randomization until the date of the study completion,an average of 3 month
  Chemotherapy delay is defined as the delay in starting the next planned chemotherapy for more than 3 days.
The duration of the chemotherapy delay in every chemotherapy cycle | From date of randomization until the date of the study completion,an average of 3 month
  The duration of the chemotherapy delay in every chemotherapy cycle
The incidence of the dose reduction | From date of randomization until the date of the study completion,an average of 3 month
  The incidence of the reduction of planned dose of chemotherapy
Relative chemotherapy dose intensity in every chemotherapy cycle | From date of randomization until the date of the study completion,an average of 3 month
  Relative chemotherapy dose intensity is defined as the actual chemotherapy dose the patient used divided by the planned chemotherapy dose,or the actual chemotherapy time divided by the planned chemotherapy time

OTHER OUTCOMES:
Incidence of adverse events | From date of randomization until the date of the study completion,an average of 3 month
  All adverse events will be recorded from the time of patients signing the informed consent form up to 30 days after the last Intervention drug is applied. the adverse event that associated with the study drug will be specially recorded.

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared by the investigators in this study